CLINICAL TRIAL: NCT07054918
Title: Isolated Positive Toxoplasma Gondii PCR in Blood
Acronym: TIPS
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: 2025 NOURRISSON (TIPS)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Toxoplasmosis
MeSH Terms: conditions — Toxoplasmosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Toxoplasmosis in immunocompromised patients is a serious, life-threatening condition that requires rapid, appropriate treatment. Diagnosis is based on PCR, notably on blood samples. Systematic blood screening is carried out for patients most at risk, to detect the disease at an early stage. Detection of parasite DNA in blood in asymptomatic patients is possible, in the absence of Toxoplasma multiplication. It has previously been proposed a distinction of two entities: toxoplasmosis disease (clinical, biological and imaging evidence of toxoplasmosis) and toxoplasmosis infection (positive PCR in the blood in the absence of clinical or radiological evidence, without progression to toxoplasmosis). Since the clinical signs of toxoplasmosis are often aspecific, a positive PCR may be the first warning result, making it difficult to determine whether the patient will progress to toxoplasmosis disease or toxoplasmosis infection.

In collaboration with the French National Reference Center for toxoplasmosis, we are proposing a retrospective multicenter study to identify possible clinical, biological or imaging criteria pointing to toxoplasmosis disease or toxoplasmosis infection as soon as the first T. gondii PCR result is positive in the blood.

ELIGIBILITY:
Inclusion Criteria:

* T. gondii positive-PCR in blood during the study period: no symptoms of toxoplasmosis since the last systematic PCR negative in blood and no history of T. gondii positive-PCR in any biological matrix for 6 weeks.

Exclusion Criteria:

* pre-analytical or analytical error leading to a false-positive result
* unknown toxoplasmosis immune status or non-immune subject
* serology in favor of acute toxoplasmosis
* congenital toxoplasmosis, ocular toxoplasmosis, toxoplasmosis in the context of HIV/AIDS
* patient opposition

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: -patient care at one of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Demographic data: age | 1 year
  expressed in years old
Demographic data: sex | 1 year
  choice between male/female
time between transplantation and positive T. gondii PCR | 1 year
  expressed in number of days
Underlying disease | 1 year
  for example: acute leukemia, solid organ transplant, ...
Ongoing anti-T. gondii prophylaxis | 1 year
  molecule name
PCR Ct value at diagnosis | 1 year
  number of cycle threshold
Outcome 1 month after first positive PCR | 1 year
  death or alive

CONTACTS AND LOCATIONS:
Overall Officials: Céline NOURRISSON, Principal Investigator — CHU de Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No